CLINICAL TRIAL: NCT04694742
Title: Ventilatory Efficiency in Critically Ill COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Ospedale Infermi Rimini (Unknown); S. Anna Hospital (Other); Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, MD, ASST Fatebenefratelli Sacco
Other Study IDs: VentRatio-19
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: ARDS
Keywords: Ventilatory ratio; Mechanical ventilation; ARDS; COVID-19; Critical illness; Dead-space
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS COVID-19: Patients who meet Berlin's ARDS diagnostic criteria, with confirmed SARS-CoV-2 infection, requiring invasive mechanical ventilation.
  Interventions: Other: data collecting

INTERVENTIONS:
Other: data collecting — Within 24h from ICU admission, the ventilatory efficiency will be assessed by the following Ventilatory Ratio equation:
  Ventilatory Ratio = [minute ventilation (ml/min) × PaCO2 (mm Hg)]/(predicted body weight × 100 × 37.5).
  Where PaCO2 is the partial pressure of carbon dioxide in mmHg in the arterial blood.
  Tha quasi-static compliance will be calculated according to the equation:
  C=Tidal Volume/(Paw plateau - PEEP total)
  where Paw plateau is the airway pressure measured during 4 seconds of inspiratory pause, PEEP total is the airway pressure measured during 4 seconds of expiratory pause.
  In the same time frame, complete blood count, d-dimer, sequential organ failure assessment score, blood gas analysis, haemodynamic and ventilatory parameters will be collected.

SUMMARY:
The new severe acute respiratory syndrome coronavirus 2019 (SARS-CoV-2) causes the illness named COVID-19, which is primarily characterized by pneumonia. As of 27 December, there have been over 79.2 million cases and over 1.7 million deaths reported since the start of the pandemic. In many cases, pneumonia evolves to acute respiratory distress syndrome (ARDS) with the need for mechanical ventilation and patient admission to intensive care unit, determining a marked increase in the need for intensive care beds worldwide.

Pulmonary involvement causes predominantly hypoxemic respiratory failure. Although COVID-19 pneumonia often falls within the diagnostic criteria of ARDS, it differs from it for some peculiar pathophysiological characteristics. In particular, patients with ARDS secondary to COVID-19 often have the compliance of the respiratory system within the normal range. A significant role in the pathophysiology of hypoxemia seems to depend on vascular alterations such as altered pulmonary vascular self-regulation, pulmonary capillary leakage, and microvascular thrombosis in a complex process known as "immunothrombosis". All together they act by altering the relationship between ventilation and perfusion and increasing the dead space, which ultimately results in impaired efficiency of the pulmonary ventilation. Among the various markers associated with the prognosis of patients with COVID-19, D-dimer is linked to both the inflammatory state and thrombotic phenomena and could help to identify patients at greater risk of developing early ventilation-perfusion changes.

This study aims at measuring the ventilatory efficiency, assessed by Ventilatory Ratio, in critically ill, mechanically ventilated, COVID-19 patients and its correlation with plasma D-dimer and quasi-static respiratory compliance.

ELIGIBILITY:
Inclusion Criteria:

All of the following:

* confirmed SARS-CoV-2 infection by RT-PCR on a nasopharyngeal swab
* severe hypoxemia due to COVID-19 who meets the diagnostic criteria of ARDS (Berlin's definition)
* invasive mechanical ventilation
* patients receiving neuromuscular blocking drugs

Exclusion Criteria:

* history of preexisting severe hypoxemia (i.e. primary pulmonary hypertension, COPD in therapy with O2 supplementation, pulmonary fibrosis, etc.)
* severe haemodynamic instability defined as:

  * Mean arterial pressure < 65 mmHg despite the infusion of norepinephrine, or epinephrine, or dobutamine, or levosimendan
  * severe left ventricular dysfunction with ejection fraction <20%
  * right ventricular failure due to pulmonary embolism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients consecutively admitted to ICU with the eligibility criteria will be enrolled in the study. They will be treated according to the standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Ventilatory ratio correlation | 24 hours from ICU admission
  Measure the correlation between ventilatory ratio, plasma D-dimer, and quasi-static compliance of the respiratory system

SECONDARY OUTCOMES:
Mortality | 30 days
  Mortality among subgroups stratified according to Ventilatory ratio and quasi-static respiratory compliance. Subgroup will be identified according centiles of the distribution values of 1) Ventilatory Ratio, and 2) quasi-static compliance both measured in the first 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Colombo, M.D., Principal Investigator — ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco
Locations (4):
- Italy (4):
  - Arcispedale Sant'Anna, Ferrara, Emilia-Romagna
  - Ospedale Infermi, Rimini, Emilia-Romagna
  - ASST Fatebenefratelli Sacco, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona, The Marches

REFERENCES:
- [Background] WHO Weekly epidemiological update - 29 December 2020 - https://www.who.int/publications/m/item/weekly-epidemiological-update---29-december-2020
- [Background] Sinha P, Calfee CS, Beitler JR, Soni N, Ho K, Matthay MA, Kallet RH. Physiologic Analysis and Clinical Performance of the Ventilatory Ratio in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2019 Feb 1;199(3):333-341. doi: 10.1164/rccm.201804-0692OC. PMID 30211618
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452